CLINICAL TRIAL: NCT05872061
Title: Senegal Market Study for Food-to-Food Fortified (F2F) Instant Porridge Flours
Acronym: SenegalMPS
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Principal Investigator / Distinguished professor, Purdue University
Other Study IDs: IRB-2021-972
Record Dates: First submitted 2023-03-13; First posted 2023-05-24 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Iron-deficiency; Vitamin A Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency; Vitamin A Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Acceptability of food-to-food fortified (FtFF) instant porridge flours — This study will evaluate the market potential of a food-to-food fortified (FtFF) flour.

SUMMARY:
The overall hypotheses is that a product designed with optimized nutritional characteristics, based on consumer preferences and leveraging local nutrient dense ingredients, can successfully deliver nutrition through sustainable market-driven approaches.

The objectives of this study were 1) to assess the nutritional adequacy of urban Senegalese households with children and 2) to determine the market potential of a locally sourced and manufactured, blended fortified, cereal-based product for the improvement of micronutrient deficiencies among children aged 24-60 months. This study simulates a market study, the investigators will conduct a product launch, determine market potential based on sales, evaluate marketing strategy to increase market share, and model the nutritional contribution of FtFF/traditionally fortified product for iron, zinc, and vitamin A. The investigators expect to provide a thorough evaluation of a business-driven strategy (for profit, social enterprise) as a sustainable tool to decrease micronutrient deficiencies.

DETAILED DESCRIPTION:
Basic design:

Participants will be approached/recruited by research assistants on the ground at designated local markets. Potential participants will be approached and consented if they agree to join the study at the time of recruitment. Research assistants will read the consent form to the participants and ensure they understand it.

Products will be produced, distributed on a weekly basis to sites. The investigators plan on introducing the "new" product to consumers at random at in-store displays at individual locations for 2 weeks, and then continue to promote (advertise) and sell the placed product for a period of 8 weeks. The following schedules are proposed:

Weeks 1-2: Product demonstrations and sampling for consumers (with promotion and free samples) Weeks 3-5: Product sold at below market cost of other millet or cereal flour products (as part of active promotion) Weeks 6-10: At one half of the locations, product sold at parity to millet or other cereal products (with advertising but no additional promotion, i.e. discount) Weeks 6-10: At one half of the locations product sold at parity +20% price to millet or other cereal products (with advertising but no additional promotion)

Data to be collected both from store managers and individual consumers. Enumerators will be trained and placed at each sales' location in the morning and evening to coincide with peak shopping times. They will be tasked with collecting a random sample of consumers who are purchasing cereals (1,200 total over 10 weeks). In this sample, both purchasers and non-purchasers of the FtFF fortified products will be identified and consented. Phone numbers will be collected and a follow up appointment/interview scheduled with half of them (600). Enumerators will also coordinate the collection of data from point of sale managers:

1. Total volume/units of FtFF fortified product sold
2. Total volume/units millet products sold
3. Total value of FtFF fortified product sold
4. TotaI value of millet product sold
5. Product comments from consumers (include any returns or complaints)
6. Number of repeat purchasers

Follow up interviews with consumers will be conducted at a private location close to the centralized market sites or points of original purchase within 2 weeks. This is to enable follow up without inconveniencing participant.

Product Production and Distribution Plan: Through a local commercial food processor Product form: 500 g size for sale. 50 g size for promotion.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age), with child(ren) 5 years of age living in the household.

Exclusion Criteria:

* No children under 5 y of age living in the household.
* Not a caregiver for the children in the household.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will collect data about dietary habits for children and the household they lived. Adult caregivers will be approached and provided the relevant information.
Sampling Method: Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Assessment of staple intake in urban Senegalese households and children | 10 weeks
  A quantitative, modified food frequency questionnaire (FFQ) will be used to assess consumption of various starch rich staples (rice, corn, sorghum, millet, potatoes, cassava) and starch-rich processed foods (bread) for the whole household and children. The caregiver will provide information about the child's amount and frequency of consumption. This will be measured in g/day*child. The investigators will ask #times/week each staple was consumed as well as the average portion size consumed each time (g).
Assessment of the nutritional adequacy of urban Senegalese households and children | 10 weeks
  Nutritional status of children in the household will be assessed using the Food Consumption Score Nutritional Quality Analysis (FCS-N) which was based on country-specific food groups. Food groups are orange fruits, orange vegetables, other fruits, eggs, dairy, organ meats, meat, fish, grains and legumes. Example of food items in the FCS-N assessment will be corroborated by a Senegalese maternal and child health expert. This will be measured in #times/week each food group was consumed.

SECONDARY OUTCOMES:
Nutritional impact of a fortified cereal-based product for the improvement of micronutrient deficiencies among children aged 24-60 months. | 10 weeks
  Fortified flour consumption will be assessed by fortified flours intake (g/child*day). Micronutrient contribution will calculated by multiplying the amount of flour consumed/child * (mg zinc/g flour), (mg iron/g flour) and (ug RAE vitamin A/g flour).

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R Hamaker, PhD, Principal Investigator — Purdue University
Locations (1):
- ITA, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: No
No PI was collected. There is not a plan to share participant information.